COMPARISON OF THE
RESULTS OF PREMATURE
BABIES STARTED
COMPLEMENTARY
FEEDING IN ADJUSTED OR
CHRONOLOGICALLY IN
THEIR SIXTH MONTH

Documented Date: June, 2 2020

Comparison of the Results of Premature Babies Started Complementary Feeding in Adjusted or Chronologically in their Sixth Month

## **Study Protocol:**

Neurological-developmental evaluations and developmental outcomes-diagnoses of premature babies are evaluated according to corrected postnatal age. Based on the limited evidence available, it can be concluded that complementary feeding may be an appropriate age for most premature babies who have reached at least the third month, generally corrected. However, for premature babies born at different gestational weeks, these periods have a relatively different meaning. A more accurate timeframe can be found in terms of complementary nutrition by evaluating chronological age and motor development together. More prospective observational studies are needed in this regard in premature babies. In the literature, there are not enough studies on the transition time to the most appropriate complementary diet for premature babies. We planned to do this prospective observational study.

Inclusion criteria for the study:

- Male / female babies who were born before the mother at the Hacettepe University Children's Hospital Neonatal Intensive Care Unit and / or Hacettepe University Adult Hospital Maternity and Birth Service and were born earlier than 37 weeks.
- Babies who are at the Hacettepe University Children's Hospital Neonatal Intensive Care Unit and / or Hacettepe University Adult Hospital Maternity and Maternity Service, were born earlier than 37 weeks and continue to be followed regularly in the neonatal outpatient clinic.
- Babies whose informed consent was obtained for their participation by the family.

Exclusion criteria:

Babies with SGA (birth weight below 10th percentile according to gestational week) by birth weight

- Babies with chromosomal anomalies
- Babies diagnosed with hypoxic ischemic encephalopathy

Babies who have had major surgical operations (gastrointestinal anomaly, severe necrotizing enterocolitis requiring surgery, major gastrointestinal system anomaly, major congenital heart anomaly, diaphragmatic hernia)

- Babies with exitus in the neonatal period
- Babies who do not continue regular polyclinic follow-up after discharge
- Babies of families who do not comply with the study protocol
- Babies with missing study data

Families who accept their babies to participate in our study will be trained with a booklet, according to the recommendations of the World Health Organization, containing the standard supplementary nutritional information we prepared beforehand.

In this study, patient groups will be randomly selected after appropriate matching. Premature babies participating in the study will be handled in three main groups (six subgroups in total).

Group 1: 29 weeks and six days of gestation and earlier

Group 2: Those whose gestational age is between 30 weeks and 33 weeks and sixth days

Group 3: Those whose gestational age is between 34 weeks and 37 weeks and sixth day

Each main group will be divided into two subgroups, according to the time to start complementary feeding (corrected sixth month or chronologically sixth month):

Group 1: 29 weeks and six days of gestation and earlier

Group 1a: complementary feeding began chronologically in the sixth month

Group 1b: Complementary feeding corrected at sixth month

Group 2: Those whose gestational age is between 30 weeks and 33 weeks and sixth days

Group 2a: complementary feeding began chronologically in the sixth month

Group 2b: complementary feeding started in the sixth month, corrected

Group 3: Those whose gestational age is between 34 weeks and 37 weeks and sixth day

Group 3a: complementary feeding began chronologically in the sixth month

Group 3b: complementary feeding started in the sixth month, corrected

Before the transition to complementary nutrition of the groups included in the study, breast milk and / or formula food, nutritional supplement (such as breast milk enhancer, protein supplement) intake will be recorded. The same polyvitamin preparation will be used for all premature babies. In accordance with the recommendation of the World Health Organization, 2 mg / kg / day standard oral iron prophylaxis will be started to all premature babies starting from the second chronological month. Immunization will be done in accordance with the national vaccination program.

The data will be added to the case report forms. In addition to routine follow-ups, families will be called on the phone monthly, information about their babies' nutrition will be asked, whether there is a problem, questions of families will be answered, and information about

complementary nutrition will be provided. At the end of the study, all data will be collected and entered into the SPSS database, which will be created.